CLINICAL TRIAL: NCT02135809
Title: Fully Covered Self Expanding Metal Stents (FCSEMS) for Refractory Pancreatic Duct Strictures in Patients With Chronic Pancreatitis
Brief Title: Pancreatic Metal Stents in Chronic Pancreatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E7093
Record Dates: First submitted 2014-05-02; First posted 2014-05-12 (Estimated); Last update posted 2019-07-09 (Actual); Status verified 2019-07

CONDITIONS: Refractory Pancreatic Duct Strictures; Painful Chronic Pancreatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FCSEMS (Experimental): Patients will receive the WallFlex Pancreatic Stent.
  Interventions: Device: WallFlex Pancreatic Stent

INTERVENTIONS:
Device: WallFlex Pancreatic Stent — Temporary placement of the WallFlex Pancreatic Stent for treatment of refractory pancreatic duct strictures in patients with painful chronic pancreatitis. Stent will be removed after 3-6 months indwell.

SUMMARY:
The purpose of this study is to document the performance of a new Fully Covered Self Expanding Metal Stents (FCSEMS) for treatment of refractory pancreatic duct strictures in patients with painful chronic pancreatitis.

DETAILED DESCRIPTION:
This study is a prospective, single arm, pre-approval study. Treatment of 10 patients will take place at 1-3 clinical centers in two phases. Phase 1 will include treatment of five patients with a three month stent indwell period at one clinical center. Phase 2 will include treatment of five additional patients with a 3-6 month stent indwell period at 1-3 clinical centers. Expected duration of participation for each patient is approximately 27 months for Phase 1 and approximately 27-30 months for Phase 2. All patients, regardless of phase, will be followed for 24 months after stent removal. Post-removal follow-up visits will occur at 1, 3, 6, 12, 18 and 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or older
2. Willing and able to comply with study procedures and follow-up schedule and provide written informed consent to participate in study
3. Chronic pancreatitis of Cremer Type IV (Segmental pancreatitis of the head of the pancreas). See Appendix for Cremer classifications.
4. Improvement of pancreatic pain during previous placement of a single pancreatic plastic stent
5. At least one of the following:

   * Abdominal pain most probably related to chronic pancreatitis
   * Recurrent dominant main pancreatic duct stricture in the head of the pancreas after prior indwell of pancreatic plastic stent(s) if pain score was available prior to preceding stent therapy. Recurrent stricture to be visually assessed at endoscopy and confirmed by recurrent main pancreatic duct dilatation at MRCP.
   * Relapsing pain due to pancreatic duct stent blockage (with only one stent in place)
6. Prior endoscopic pancreatic sphincterotomy (EPS), historically or to be provided at time of SEMS placement with informed patient consent.

Exclusion Criteria:

1. Strictures caused by malignancies
2. Biliary strictures caused by chronic pancreatitis
3. Perforated duct.
4. Ansa pancreatica or H anatomy
5. Pancreatic duct stenoses not located in the head of the pancreas
6. Failed access during an attempted ERCP on a prior date
7. Prior pancreatic metal stent(s)
8. Concurrent ESWL (Extracorporeal Shock Wave Lithotripsy) during the same treatment session
9. Patients for whom endoscopic techniques are contraindicated.
10. Patients who are currently enrolled in another investigational study that would directly interfere with the current study, without prior written approval from the sponsor
11. Inability or refusal to comply with the follow-up schedule including subject living at such a distance from the investigational center that

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2017-03-30 (Actual)

PRIMARY OUTCOMES:
Decrease of pain caused by refractory benign pancreatic duct strictures secondary to chronic pancreatitis | 3 months after study stent removal
  Clinical success defined as decrease of pain caused by refractory benign pancreatic duct strictures secondary to chronic pancreatitis 3 months after stent removal compared to baseline prior to stent indwell period.

SECONDARY OUTCOMES:
Occurrence and severity of serious adverse events related to the stenting procedure, to the indwelling stent and/or to stent removal | Duration of study participation, an average of 27-30 months
Stent placement success | Study Stent Placement Procedure
  Ability to deploy the stent in satisfactory position (Stent Placement Success). Satisfactory position is defined as the stent being across the stricture, without visible impaction at an angle and distal end visible into the duodenum.
Type of additional intervention within pancreatic duct | Duration of study participation, an average of 27-30 months
Stent removal success | Study Stent Removal
  Successful stent removal (Stent Removal Success) defined as ability to remove stent endoscopically (grasper, snare, stent-in-stent) without serious stent removal-related adverse events
Change of pain medication intake | Duration of study participation, an average of 27-30 months
  Change of pain medication intake (type of medication) from baseline to each follow-up visit.
Number of device events | Duration of study participation, an average of 27-30 months
  Device Events, including findings not associated with adverse events, such as but not limited to asymptomatic stent migration.
Stricture resolution of pancreatic duct after stent removal | Study Stent Removal
  Assessment of pancreatic duct after stent removal compared to baseline, including ERCP to document extent of stricture resolution, extent of resolution of ductal dilation above the treated dominant stricture, and presence or absence of secondary ductal strictures at the level of where the proximal edge of the stent was located
For patients who proceed to surgery, impact of prior SEMS on surgical outcomes. | Up to surgery
Stent functionality | Up to time of study stent removal,average of 3-6 months on study
  Stent functionality: Relief of pain caused by refractory benign pancreatic duct strictures secondary to chronic pancreatitis at 3 days, 2 weeks, 1 month, 2 months, 4 months (Phase 2 patients as applicable) and just prior to stent removal compared to baseline prior to stent placement, using established pancreatic pain score
Stricture Resolution at stent removal | Study Stent Removal
  Stricture Resolution at stent removal, defined as pancreatographic confirmation of drainage of injected contrast medium after stent removal without visible persistent stricture
Time to Recurrence of Stricture | Duration of study participation, an average of 27-30 months
  Time to Recurrence of Stricture, established in patients who had stricture resolution at stent removal and defined as time elapsed from stent removal till recurrence of pain with associated documentation of narrowing of pancreatic duct. Recurrence of stricture will be documented at the time it is identified and absence of stricture recurrence will be ascertained at 1, 3, 6, 12, 18 and 24 months after stent removal. Pain will be documented using an established pancreatic pain score.
Reason for additional intervention within pancreatic duct | Duration of study participation, an average of 27-30 months
Timing of additional intervention within pancreatic duct | Duration of study participation, an average of 27-30 months

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Devière, MD, PhD, Principal Investigator — ULB Erasme Hospital
Locations (1):
- ULB Erasme Hospital, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No